CLINICAL TRIAL: NCT07204184
Title: Cervical and Lumbosacral Transspinal Stimulation to Reconnect the Injured Human Spinal Cord
Brief Title: Multisite Transspinal Stimulation for Augmenting Recovery in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Knikou, PT, MBA, PhD (Other)
Responsible Party: Sponsor-Investigator, Maria Knikou, PT, MBA, PhD, Professor, Senior Research Scientist, City University of New York
Organization: City University of New York (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: C41217GM; C41217GM (Other Grant/Funding Number: NYSDOH, SCIRB)
Record Dates: First submitted 2025-09-10; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries (Complete and Incomplete)
Keywords: transspinal stimulation; robotic gait training; locomotor training; non-invasive; multi-modal rehabilitation; clinical biomarkers; neurophysiological biomarkers; sensorimotor recovery
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers who will perform data reduction, data analysis and statistical analysis of the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Multisite transspinal stimulation at rest (Active Comparator): Cervical and lumbosacral non-invasive transspinal tonic stimulation will be delivered at 30 Hz frequency (charge-balanced, symmetric, biphasic rectangular pulses of a 1-ms width per phase) at paresthesia levels or higher depending on each participant's comfort level while participants rest lying on the back. A total of 20 sessions (weekdays excluding weekends and holidays), each for 1 hour, will be administered.
  Interventions: Device: Multisite transspinal stimulation at rest
- Multisite transspinal stimulation during robotic gait training (Active Comparator): The investigators will deliver cervical and lumbosacral non-invasive transspinal tonic stimulation at 30 Hz frequency (charge-balanced, symmetric, biphasic rectangular pulses of a 1-ms width per phase) at paresthesia levels or higher depending on each participant's comfort level during assisted stepping with the Lokomat 6 Pro, a robotic device that helps the legs step and provides as needed body weight support. A total of 20 sessions (weekdays excluding weekends and holidays), each for 1 hour, will be administered.
  Interventions: Device: Multisite transspinal stimulation during robotic gait training

INTERVENTIONS:
Device: Multisite transspinal stimulation at rest — The intervention, combined cervical and lumbar transspinal stimulation, will be used for the first time to reconnect the spared neuronal pathways of the injured human spinal cord. The intervention will be administered while at rest lying on the back or during robotic gait training. Cervical and lumbar transspinal stimulation will be delivered via surface active electrodes placed on the back of the neck and on low back, and four returning electrodes placed on each clavicle and iliac crest.
  Other Names: transcutaneous spinal cord stimulation; transspinal stimulation; robotic gait training; locomotor training; non-invasive spinal cord stimulation
  Arms: Multisite transspinal stimulation at rest
Device: Multisite transspinal stimulation during robotic gait training — The intervention, combined cervical and lumbar transspinal stimulation, will be administered during robotic gait training. Cervical and lumbar transspinal stimulation will be delivered via surface active electrodes placed on the back of the neck and on low back, and four returning electrodes placed on each clavicle and iliac crest while participants step with the help of the Lokomat 6 Pro, a robotic device that helps the legs step. Locomotor training will depend on the ability of each participant to step without foot dragging. Over the training course, we will adjust the body weight support, ankle straps position, and leg guidance force. The tension of the ankle straps will be adjusted based on the right and left tibialis anterior muscle strength evaluated every 2 weeks. Body weight support and leg guidance force will be adjusted based on presence or absence of knee buckling during standing.
  Other Names: locomotor training; body weight supported assisted step training
  Arms: Multisite transspinal stimulation during robotic gait training

SUMMARY:
A well-established rehabilitation strategy for improvements of standing and walking ability in persons with spinal cord injury (SCI) is step training on a motorized treadmill with body weight support. A promising intervention is stimulation of the spinal cord through the skin (transspinal). No single intervention is likely to significantly improve long-term function after SCI on its own. Rather, combinatorial treatments that work synergistically and can be used at different clinical settings is the answer to target recovery in people with SCI. The objective of this clinical trial is to develop a non-invasive combinatorial intervention that can be used worldwide in different clinical settings. The investigators will use cervical and lumbosacral transspinal stimulation to augment the benefits of locomotor training and affect vital body functions after SCI. The investigators will deliver non-invasive cervical and lumbosacral transspinal stimulation alone or with step training to improve upright posture, walking, bladder, sex, and bowel function in persons with incomplete SCI. The noninvasive nature of the intervention holds minimal risk that outweighs the benefits.

DETAILED DESCRIPTION:
The main objective of this hypothesis-based and need-driven clinical research trial is to develop novel rehabilitation strategies and impact clinical practice and care for people with spinal cord injury (SCI). The investigators will use non-invasive transspinal stimulation over the cervical and lumbosacral enlargements, the spinal location of arm and leg motor circuits, to augment the benefits of locomotor training and improve recovery of standing and walking ability in individuals with SCI. This trial is a pilot (or small-scale) clinical trial on cervical and lumbosacral transspinal stimulation administered alone at rest or during assisted step training in people with SCI to establish safety and efficacy.

The investigators' specific aims are as follows:

1. Determine the underlying physiological actions of paired cervical and lumbosacral transspinal stimulation in people with and without SCI. To address Specific Aim 1, in 12 people with incomplete SCI (AIS B, C, D) and 12 healthy control subjects (age and gender match) we will establish the effects of a) cervical transspinal stimulation on soleus H-reflexes and leg transspinal evoked potentials (TEPs), and the effects of lumbosacral transspinal stimulation on flexor carpi radialis (FCR) H-reflexes, and arm TEPs at rest; and b) the effects of cervical and lumbosacral paired transspinal stimulation on joint coordination and muscle synergies during walking on a motorized treadmill (healthy controls) or with a robotic gait system training (Lokomat) in participants with SCI.
2. Determine if cervical and lumbosacral transspinal stimulation reconnects the injured human spinal cord, strengthens the weak remnant neuronal pathways, and augments the benefits of locomotor training. To address Specific Aim 2, a total of 24 people with incomplete SCI (AIS B, C, D) will be enrolled. Half will receive cervical and lumbosacral transspinal stimulation at rest. The other half of participants will receive cervical and lumbosacral transspinal stimulation during assisted stepping with a robotic gait system (Lokomat 6 Pro®).

Both groups will receive 20 sessions (5 sessions/week) of 1-hr duration each. Cervical and lumbosacral transspinal stimulation will be delivered at 30 Hz at or above paresthesia intensities based on each participant's comfort levels. For both groups, the investigators will establish safety based on adverse events, and efficacy based on clinical assessments and neurophysiological biomarkers. Before and after the intervention the investigators will 1) establish changes in non-somatic vital bladder, bowel, and sexual body functions, 2) perform clinical assessments of spasticity, standing and walking ability, and 3) perform state-of-the-art experiments to establish changes in neurophysiological biomarkers.

The investigators will use neurophysiological biomarkers to probe actions of the proposed intervention (cervical and lumbosacral transspinal stimulation), use combination of interventions, and address safety and efficacy of intervention via adverse events and neurophysiological biomarkers. Furthermore, the investigators will 1) identify and validate biomarkers for diagnosis, prognosis, and evaluation of treatment efficacies, and 2) maximize the function of the residual neural circuitry, including harnessing neuroplasticity and recovery to improve function after SCI.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to comply with all study procedures and availability for the duration of the study.
* Ability to understand the consent form and sign the consent form.
* In good general health as evidenced by medical history.
* Diagnosed with incomplete SCI (AIS B, C, D).
* Bone mineral density of the hip (proximal femur) T-score <3.5 SD from age- and gender-matched normative data.
* Lesion above thoracic (T) 10 to ensure absent lower motoneuron lesion.
* The presence of soleus and FCR H-reflexes.
* Absent permanent ankle joint contractures prevent passive or active ankle movement because corticospinal and spinal excitability is based on the ankle angle. The ankle straps of the Lokomat also require flexible ankle joints.
* A diagnosis of first time SCI due to trauma, vascular, or orthopedic pathology.
* Time after SCI of more than 6 months.
* Stable medical condition without cardiopulmonary disease or cognitive impairment.

Exclusion Criteria:

* Supraspinal lesions.
* Neuropathies of the peripheral nervous system.
* Significant degenerative neurological disorders of the spine or spinal cord.
* Diagnosed with AIS A.
* Presence of pressure sores.
* Advanced urinary tract infection.
* Neoplastic or vascular disorders of the spine or spinal cord.
* Participation in an ongoing research study or new rehabilitation program.
* Pregnant women or women who suspect they may be or may become pregnant will be excluded from participation because the risks of thoracolumbar stimulation to the fetus are unknown.
* People with cochlear implants, pacemakers, implanted infusion device, and/or implanted stimulators of any type and purpose will be excluded to avoid their malfunction due to stimulation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Soleus H-reflex recruitment curve | Before and 1 day after all intervention sessions are completed.
  Investigators will deliver single pulses of 1 ms duration every 5 seconds at increasing intensities to the posterior tibial nerve behind the knee to assemble the soleus H-reflex recruitment curve. At least 50 responses will be recorded. From the recruitment curve, the investigators will estimate changes in the slope and stimulation intensities for reflex threshold.
Soleus H-reflex rate-dependent depression | Before and 1 day after all intervention sessions are completed.
  Soleus H-reflexes following posterior tibial nerve of the right leg behind the knee with a 1-ms pulse randomly at 1, 3, 5, 8, and 10 s inter-pulse intervals will be recorded. At each inter-pulse interval, 15 responses will be recorded. Stimulation will be delivered via a ball shape electrode and responses will be recorded from leg muscles with surface electrodes. The smaller the soleus H-reflex amplitude when evoked every 1 second the larger the spinal inhibition. Recovery of spinal inhibition will be considered when the soleus H-reflex depression at 1 second is statistically significant different before and after the intervention.
Soleus H-reflex phase-dependent modulation during stepping | Before and 1 day after all intervention sessions are completed.
  Each participant will step with the assistance of the Lokomat, and the investigators will record soleus H-reflexes randomly across 16 equal time bins into which each step cycle is divided. The posterior tibial nerve behind the knee will be stimulated at motor threshold. Stimulations will be triggered based on the foot switch signal. Under physiological conditions, the soleus H-reflex during walking largely is facilitated during the stance phase and inhibited during the swing phase. Recovery of spinal locomotor circuits will be based on the amplitude of the soleus H-reflex during the stance and swing phases of gait, and how much is facilitated and inhibited during the stance and swing phases after intervention compared to before intervention for each participant.
Leg transspinal evoked potentials recruitment curves | Before and 1 day after all intervention sessions are completed.
  The investigators will deliver single 1 ms pulses every 5 seconds at increasing intensities with a surface electrode to the low back to assemble the recruitment curves of transspinal evoked potentials recorded from leg muscles with surface electrodes. Participants will lay on their back on a treatment table. From the recruitment curve, the slope and excitation threshold will be established and the intervention will be considered effective when statistical significant differences on their amplitude between before and after values is established.
Flexor carpus radialis H-reflex recruitment curve | Before and 2 days after all intervention sessions are completed.
  The investigators will stimulate the median nerve with a bipolar surface electrode at the elbow with single 1-ms pulses at increasing intensities every 5 seconds while participants are seated. At least 50 responses will be recorded. From the recruitment curve, the slope and excitation threshold will be established. The intervention will be considered effective when statistical significant differences between before and after values is found.
Flexor carpus radialis H-reflex rate dependent depression | Before and 2 days after all intervention sessions are completed.
  Flexor carpus radialis H-reflexes following median nerve stimulation with a surface bipolar electrode of the right arm at the elbow with a 1-ms pulse will be recorded randomly at 1, 3, 5, 8, and 10 s inter-pulse intervals. At each inter-pulse interval, 15 responses will be recorded. Responses will be recorded from arm muscles with surface electrodes. Under physiological conditions, the reflex is smaller when evoked every 1 second compared to that evoked every 10 seconds. Recovery of spinal inhibition will be considered when a smaller reflex is evoked every 1 second after the intervention compared to that observed before intervention.
Arm transspinal evoked potentials recruitment curves | Before and 2 days after all intervention sessions are completed.
  The investigators will deliver single 1 ms pulses every 5 seconds at increasing intensities to the back of the neck with a surface electrode to assemble the recruitment curves of transspinal evoked potentials recorded from arm muscles with surface electrodes. Participants will lay on their back on a treatment table. From the recruitment curve, the slope and excitation threshold will be established and the intervention will be considered effective when statistical significant differences between before and after intervention is established.

SECONDARY OUTCOMES:
2-Minute Walk Test | Before and 1-day after all intervention sessions are completed.
  The 2-Minute Walk Test is a physical assessment measuring aerobic capacity and endurance. Participants will walk with or without assistive devices as far as possible for two minutes in a hallway. The total distance walked is recorded, and will be compared to normative values for the participant's age and gender to identify potential limitations or track progress over time.
  There is currently no single established Minimal Clinically Important Difference for the 2-minute walk test in people with spinal cord injury. However, a recent study showed that in the subacute phase of rehabilitation a 2-Minute Walk Test Minimal Clinically Important Difference is considered when the increase is 31 meters. However, other research studies indicate that the Minimal Clinically Important Difference can vary significantly depending on the specific patient population, rehabilitation stage, disability level, and age.
10-Meter Walk Test | Before and 1-day after all intervention sessions are completed.
  The 10-Meter Walk Test is a performance measure and assesses the walking speed in meters per second over a short duration. Participants will walk 10 meters and the time needed to cover the 10 meters will be recorded. The minimal clinically important difference for the 10-meter walk test in spinal cord injury is approximately 0.13 m/s, a value established for individuals with incomplete SCI within one year of injury. This means that recovery of walking ability will be based on when the speed is improved by 0.13 m/s.
Sexual function | Before and 1-day after completion of all intervention sessions.
  Participants will complete a brief questionnaire on sexual function before and after intervention. The questionnaire is the International Spinal Cord Injury sexual function for male and female. The answers to the questions include: normal, reduced/altered, absent, and unknown/not applicable. Improvement from the intervention will be considered when more "normal" answers replace the "reduced-absent or absent" answers.
Bladder function | Before and 1-day after completion of all intervention sessions.
  The Overactive Bladder Symptom Score (OABSS) questionnaire will be answered by the participants before and after intervention to establish recovery or changes of the bladder function. The maximum score is 15 and the minimum score is 0. The smaller the score the better the outcome.
Bowel function | Before and 1-day after all intervention sessions are completed.
  The University of Michigan Spinal Cord Injury Model Systems for Bowel function questionnaire will be used to establish recovery or changes. The answers are descriptive including yes or no or at least daily or never. A number 1 will be given to the answer that represents the least impact of bowel function on the quality of life and satisfaction. When the sum of scores is lower by at least 20% after the intervention, it will be regarded as improvements in bowel function.
Modified Ashworth Scale | Before and 1-day after all interventions are completed.
  The Modified Ashworth Scale assesses spasticity in the lower extremity. The investigators will apply a quick manual stretch to the ankle. A score from 0 to 4 will be given, where 0 indicates no increase in tone and 4 signifies complete rigidity. A score of 1 or 1+ indicates a slight increase in tone with a catch, while 2 means a marked increase, and 3 signifies a considerable increase that makes passive movement difficult. The maximum score is 4 and the minimum score is 0. The lower the score the better the outcome or recovery. A minimal clinically important difference for the Modified Ashworth Scale is 0.45 for the lower extremity.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA KNIKOU, PT, MBA, PhD, Principal Investigator — City University of New York, College of Staten Island
Locations (1):
- College of Staten Island (Building 5N-218), Staten Island, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited Individual participant data (IPD) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Study Protocol and Statistical Analysis Plan (SAP) will be shared at the completion of the clinical trial.
Access Criteria: IBD and supporting information will be available to the investigators of the clinical trial, institutional review board (IRB) committees, and the funder. IBD and supporting information will be available to other researchers upon completion and publication of the results of the clinical trial upon written request to the Principal Investigator.
  The investigators of the clinical trial, institutional review board (IRB) committees, and the funder will have access to coded muscle activity and compound muscle action potentials stored as Spike 2 or LabView data files in a password-protected computer, as well as information entered in handwriting in experimental forms. Clinical research evaluation tests are logged in a printed document and saved in a locked file cabinet separate from medical records and signed consent forms. All data, digital or written in forms, are saved with the code given to each participant

REFERENCES:
- [Background] Knikou M, Mummidisetty CK. Locomotor training improves premotoneuronal control after chronic spinal cord injury. J Neurophysiol. 2014 Jun 1;111(11):2264-75. doi: 10.1152/jn.00871.2013. Epub 2014 Mar 5. PMID 24598526
- [Background] Smith AC, Rymer WZ, Knikou M. Locomotor training modifies soleus monosynaptic motoneuron responses in human spinal cord injury. Exp Brain Res. 2015 Jan;233(1):89-103. doi: 10.1007/s00221-014-4094-7. Epub 2014 Sep 10. PMID 25205562
- [Background] Knikou M, Smith AC, Mummidisetty CK. Locomotor training improves reciprocal and nonreciprocal inhibitory control of soleus motoneurons in human spinal cord injury. J Neurophysiol. 2015 Apr 1;113(7):2447-60. doi: 10.1152/jn.00872.2014. Epub 2015 Jan 21. PMID 25609110
- [Background] Murray LM, Knikou M. Remodeling Brain Activity by Repetitive Cervicothoracic Transspinal Stimulation after Human Spinal Cord Injury. Front Neurol. 2017 Feb 20;8:50. doi: 10.3389/fneur.2017.00050. eCollection 2017. PMID 28265259
- [Background] Islam MA, Pulverenti TS, Knikou M. Neuronal Actions of Transspinal Stimulation on Locomotor Networks and Reflex Excitability During Walking in Humans With and Without Spinal Cord Injury. Front Hum Neurosci. 2021 Feb 18;15:620414. doi: 10.3389/fnhum.2021.620414. eCollection 2021. PMID 33679347
- [Background] Zaaya M, Pulverenti TS, Knikou M. Transspinal stimulation and step training alter function of spinal networks in complete spinal cord injury. Spinal Cord Ser Cases. 2021 Jul 3;7(1):55. doi: 10.1038/s41394-021-00421-6. PMID 34218255
- [Background] Sayed Ahmad AM, Zaaya M, Harel NY, Knikou M. Transspinal stimulation preceding assisted step training reorganizes neuronal excitability and function of inhibitory networks in spinal cord injury: A randomized controlled trial. medRxiv [Preprint]. 2025 Jun 12:2025.06.11.25329338. doi: 10.1101/2025.06.11.25329338. PMID 40585100
- [Background] Knikou M, Murray LM. Repeated transspinal stimulation decreases soleus H-reflex excitability and restores spinal inhibition in human spinal cord injury. PLoS One. 2019 Sep 26;14(9):e0223135. doi: 10.1371/journal.pone.0223135. eCollection 2019. PMID 31557238
- [Background] Sayed Ahmad AM, Skiadopoulos A, Knikou M. Interactions between arm and leg neuronal circuits following paired cervical and lumbosacral transspinal stimulation in healthy humans. Exp Brain Res. 2024 Sep;242(9):2229-2239. doi: 10.1007/s00221-024-06891-y. Epub 2024 Jul 22. PMID 39034329

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-09-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT07204184/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT07204184/ICF_001.pdf